CLINICAL TRIAL: NCT04046107
Title: Safety and Immunotherapeutic Activity of Cemiplimab in Participants With HBV on Suppressive Antiviral Therapy: A Phase I/II Ascending Multiple Dose Study
Brief Title: Safety and Immunotherapeutic Activity of Cemiplimab in Participants With HBV on Suppressive Antiviral Therapy
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Temporarily closed to enrollment
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5368; 38410 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Hepatitis B Virus
Keywords: Hepatitis B; Chronic hepatitis B; Functional cure; Immunotherapy; Checkpoint inhibitor therapy
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Cemiplimab (0.3 mg/kg) (Experimental): Participants will receive cemiplimab 0.3 mg/kg dosed in two infusions, one infusion at Week 6 and Week 12.
  Interventions: Biological: Cemiplimab
- Cohort 2: Cemiplimab (1 mg/kg) (Experimental): Participants will receive cemiplimab 1 mg/kg dosed in two infusions, one infusion at Week 6 and Week 12.
  Interventions: Biological: Cemiplimab
- Cohort 3: Cemiplimab (3 mg/kg) (Experimental): Participants will receive cemiplimab 3 mg/kg dosed in two infusions, one infusion at Week 6 and Week 12.
  Interventions: Biological: Cemiplimab

INTERVENTIONS:
Biological: Cemiplimab — Administered as an intravenous (IV) infusion
  Other Names: REGN2810

SUMMARY:
The purpose of this study is to evaluate the safety and immunotherapeutic activity of cemiplimab in participants with hepatitis B virus (HBV) on suppressive antiviral therapy.

DETAILED DESCRIPTION:
The study consists of up to three cemiplimab dose cohorts (n=10 participants each). The cohorts will open sequentially, based on the safety of the previous cohort. Cohort 1 will open first to examine the lowest dose. When Cohort 1 participants have completed study week 18 visit and there are no safety concerns, Cohort 2 will open for enrollment. A similar assessment will be conducted with Cohort 2 to make a decision on opening Cohort 3. In each cohort, participants enter the study 6 weeks prior to initiation of treatment. The 6-week lead-in period is followed by a 6-week treatment period where two infusions of cemiplimab are administered 6 weeks apart, at study weeks 6 and 12.

The total study duration per participant is 90 weeks, including 78 weeks of follow-up after the treatment period. Study visit schedule includes visits at entry, and weeks 6, 7, 8, 10, 12, 13, 14, 16, 17, 18, 22, 24, 30, 36, 54, 72 and 90. Evaluations include: a medical and medication history; assessment of HBV antiviral therapy adherence; physical exam; blood, urine, and fecal collection; rectal swab; liver biopsy and fine needle aspiration; and optional leukapheresis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HBV infection (defined as hepatitis B surface antigen [HBsAg] positive).
* Receiving treatment at the time of study entry and for ≥12 months prior to study entry with HBV-active nucleos(t)ides, with tenofovir- or entecavir-containing therapy: tenofovir disoproxil fumarate (TDF), tenofovir alafenamide (TAF), TDF/emtricitabine (FTC), TAF/FTC, or entecavir.
* Ability and willingness of participant to provide informed consent.
* Ability and willingness of participant to continue HBV antiviral therapy throughout the study.
* Weight ≥40 kg and <200 kg.
* Evidence of limited or no evidence of fibrosis (F0-F2) by liver biopsy or non-invasive alternative, as defined in the study protocol.
* The following laboratory values obtained within 60 days prior to study entry:

  * HBV DNA level <20 IU/mL
  * Documentation of hepatitis B e antigen (HBeAg) status (positive or negative)
  * Hemoglobin ≥14.0 g/dL for male, ≥12.0 g/dL for female participants
  * Platelets ≥150,000/mm^3
  * Absolute neutrophil count (ANC) >1500/mm^3
  * International normalized ratio (INR) ≤1.1
  * Albumin ≥3.5 g/dL
  * Creatinine Clearance ≥60 mL/min, as calculated by the Cockcroft-Gault equation

    * NOTE: A calculator for the Cockcroft-Gault equation is available on the Data Management Center (DMC) website at www.fstrf.org.
  * Aspartate aminotransferase (AST) serum glutamic:oxaloacetic transaminase (SGOT) <1.25 x ULN
  * ALT serum glutamic:pyruvic transaminase (SGPT) <1.25 x ULN
  * Direct bilirubin ≤1.0 x ULN
  * AM cortisol >10 mcg/dL and <ULN

    * NOTE A: Female participants on estrogen-containing oral contraception or other exogenous estrogen treatment may repeat the AM cortisol as part of screening to determine eligibility. AM cortisol should be drawn prior to 12 noon or per local lab requirements.
    * NOTE B: Participants with a low cortisol level that was drawn after 10:00 AM may repeat the AM cortisol as part of screening to determine eligibility.
  * Normal creatinine phosphokinase (CPK) level
  * Thyroid stimulating hormone (TSH) and free thyroxine (T4) level within normal limits
  * Fasting blood glucose <126 mg/dL
* Interferon-gamma release assay (IGRA) for tuberculosis (TB) with negative results within 90 days prior to study entry, OR prior positive TB IGRA or positive purified protein derivative (PPD) skin test with documented evidence of completed prophylaxis treatment.
* HCV antibody negative result within one year prior to study entry; or if the participant is HCV antibody positive, an unquantifiable HCV RNA result (< lower limit of quantification [LLOQ], either target detected, or target not detected) within 60 days prior to study entry.
* Documentation of completion of SARS-CoV-2 vaccine series and up-to-date additional or booster immunizations, as recommended by local country guidance
* Participants of reproductive potential, a negative urine or serum pregnancy test at screening, and again within 48 hours prior to study entry by any US clinic or laboratory that has CLIA certification or its equivalent, or is using a point of care (POC)/ CLIA-waived test, or at any Network-approved non-US laboratory or clinic that operates in accordance with GCLP and participates in appropriate EQA programs
* All participants must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, oocyte donation, in vitro fertilization).
* When participating in sexual activity that could lead to pregnancy, participants must agree to use at least two reliable forms of contraceptive simultaneously, over the time period of 36 weeks following study entry (to include time period up to 6 months after last infusion). Such methods include:

  * Condoms (male or female) with or without a spermicidal agent
  * Diaphragm or cervical cap with spermicide
  * Intrauterine device (IUD)
  * Tubal ligation
  * Hormone-based contraceptive

    * NOTE: Providers and participants should be advised that not all contraceptive choices listed above can prevent HBV transmission. Study participants who are sexually active with HBV negative or unknown HBV serostatus partners should be advised that they need to consider effective strategies to reduce the risk of HBV transmission and meet the requirement for effective contraception during their participation in the study. Study participants should discuss contraceptive choices and HBV risk-reduction methods with their health care provider.
* Participants who are not of reproductive potential (women who have been post-menopausal for at least 24 consecutive months or have undergone hysterectomy and/or bilateral oophorectomy or salpingectomy or men who have documented azoospermia) are eligible without requiring the use of contraceptives. Acceptable documentation of menopause or sterilization is specified below.

  * Written or oral documentation communicated by clinician or clinician's staff of one of the following:

    * Physician report/letter
    * Operative report or other source documentation in the patient record (a laboratory report of azoospermia is required to document successful vasectomy)
    * Discharge summary
    * Follicle stimulating hormone-release factor (FSH) measurement elevated into the menopausal range as established by the reporting laboratory
* Intention to comply with the dosing instructions for study drug administration and ability to complete the study schedule of assessments.

Exclusion Criteria

* Any malignancy within the 5 years prior to study entry or current malignancy requiring cytotoxic therapy.

  * NOTE: A history of non-melanoma skin cancer (e.g., basal cell carcinoma or squamous cell skin cancer) at any time is not exclusionary.
* Current chronic, acute, or recurrent bacterial, fungal, or viral (other than HBV) infections that are serious, in the opinion of the site investigator, and that required systemic therapy within 30 days prior to study entry.
* Prior history of or active autoimmune disorders including but not limited to inflammatory bowel diseases, scleroderma, severe psoriasis, myocarditis, uveitis, pneumonitis, systemic lupus erythematosus, rheumatoid arthritis, optic neuritis, myasthenia gravis, adrenal insufficiency, hypothyroidism and/or hyperthyroidism, autoimmune thyroiditis, hypophysitis, multiple sclerosis, or sarcoidosis.

  * NOTE: For questions related to the definition of autoimmune disorders, sites should contact the team per the study protocol.
* Any known acquired or congenital immune deficiency.
* History of chronic obstructive pulmonary disease (COPD).
* History of significant pulmonary conditions.
* Unstable asthma (e.g., sudden acute attacks occurring without an obvious trigger) or asthma requiring:

  * Daily steroid or long-acting beta-agonist prevention
  * Hospitalization in the 2 years prior to entry
* A history of chronic congestive heart failure or other significant cardiac condition.
* Any active clinically significant medical condition that, in the opinion of the site investigator, would place the participant at increased risk.
* History of non-infectious pneumonitis within the last 5 years prior to study entry.
* Retinopathy or uveitis within 180 days prior to study entry.
* Any acute or chronic psychiatric diagnoses that, in the opinion of the investigator, make the participant ineligible for participation.
* Any vaccination within 30 days prior to entry with the exception of SARS-CoV-2 vaccination..

  * NOTE: Individuals who require vaccination must delay screening for the study until 30 days after receiving the last injection.
* Human immunodeficiency virus (HIV) infection.
* Evidence of current (within 1 year prior to entry) Hepatitis delta virus (HDV) infection (HDV antibody positive).
* Acute or serious illness, in the opinion of the site investigator, requiring systemic treatment and/or hospitalization within 30 days prior to study entry.
* Alpha-Fetoprotein (AFP) >100 within 60 days prior to study entry in the absence of imaging within the prior 6 months prior to study entry to exclude hepatocellular carcinoma (HCC).
* Any known bleeding disorder (i.e., hemophilia).
* Receipt of investigational drug or device within 6 months prior to study entry.
* History of treatment with a phosphoinositide 3-kinase inhibitor, including idelalisib.
* History of checkpoint inhibitor treatment including anti-programmed death-1 (anti-PD-1), anti-programmed death-ligand 1 (anti-PD-L1) or anti-cytotoxic T-lymphocyte antigen 4 (anti-CTLA-4) antibodies.
* History of immunoglobulin IgG therapy.
* Receipt of interferon (IFN) therapy within 12 months prior to study entry.
* Use of immunomodulators (e.g., interleukins, cyclosporine), systemic cytotoxic chemotherapy, or corticosteroid therapy.

  * NOTE A: Participants receiving topical corticosteroids will not be excluded.
  * NOTE B: Participants receiving inhaled corticosteroids will be excluded.
* Intent to use immunomodulators (e.g., IL-2, IL-12, interferon [IFNs], or TNF modifiers) or corticosteroids (other than topical steroids) during the course of the study.
* Current HCV antiviral therapy or receipt of HCV treatment in the 6 months prior to study entry.
* Use of anticoagulants within the 30 days prior to study entry.
* Prior treatment with other immune modulating agents that was associated with toxicity that resulted in discontinuation of the immune-modulating agent.
* Current use or intent to use biotin ≥5 mg/day, including within dietary supplements during the study.

  * NOTE: Please see the study protocol for a list of other names used for biotin that should be looked for on the labels of dietary supplements.
* Positive thyroid peroxidase (TPO) antibody result within 60 days prior to study entry.
* Positive glutamic acid decarboxylase antibody (GAD65 Ab) result within 60 days prior to study entry.
* Positive islet cell antibody result within 60 days prior to study entry.
* Positive antinuclear antibody (ANA) ≥1:80 within 60 days prior to study entry.
* Anti-smooth muscle antibody >1:80 within 60 days prior to study entry.
* Immunoglobulin G (IgG) ≥1.2 x ULN within 60 days prior to study entry.
* Known allergy/sensitivity or any hypersensitivity to components of cemiplimab (anti-PD-1) or its formulation or previous mAb treatments.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Breastfeeding or pregnancy.
* A male participant with a pregnant female sexual partner.
* For participants in the optional leukapheresis (LA) component, prior history of difficulty establishing venous access or current contraindication for LA, in the opinion of the site investigator and based on pre-LA assessments listed in the study protocol.

  * NOTE: Participants unwilling or unable to complete LA are still eligible for enrollment into the main study.
* Participants with a history of solid organ transplant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experienced any targeted safety event that is related to study treatment | From Week 6 to Week 18
  Targeted safety events include:
  * Hepatic encephalopathy
  * Ascites
  * Grade 2 or higher ALT elevation with INR greater than 1.5 or direct bilirubin greater than 1.5, unless occurring as part of HBeAg or HBsAg seroconversion to anti-HBe or anti-HBs or greater than 1 log decline in quantitative HBsAg with ALT resolution to Grade 1 or less within 60 days of elevation.
  * Non-hepatic AE of Grade 3 or higher
  * Adrenal insufficiency or adrenal crisis, confirmed, Grades 1-3
  * Myocarditis, Grades 1-3
  * Pneumonitis, Grades 2-3
  * Infusion-related reaction, Grade 3
  * Rash, Grade 3
  * Uveitis, Grades 1-3
  * Immune mediated hyper- or hypothyroidism, Grades 2-3
  * Colitis, Grade 3 or higher
  * Myositis, Grades 2-3
  * Immune-mediated hepatitis
  * Death
  DAIDS AE Grading Table (V2.1) is used.
Number of participants who discontinue treatment and/or study which is related to any adverse event | From Week 6 to Week 18
  Attributed to any adverse event as reported by the site
Number of participants with any AE | From entry to Week 90
  Study protocol requires reporting of all targeted events (listed in Primary Outcome Measure 1 above), all Grade 1 or higher AEs, and any AE that occurs during the infusion or within 24 hours after infusion. DAIDS AE Grading Table (V2.1) is used.

SECONDARY OUTCOMES:
Change in quantitative HBsAg from pre-treatment | Entry and Weeks 6, 8, 12, 14, 18, 24, 36, 54, 72, 90
  Pre-treatment value is the average of measurements at study entry and treatment initiation
Number of participants with detectable HBsAg | Entry and Weeks 6, 12, 18, 36, 54, 72, Week 90
  HBsAg detections based on the qualitative assay
Number of participants with anti-HBs conversion from negative (at study Week 6) to positive at a subsequent visit | Weeks 6, 12, 18, 36, 54, 72, 90
  Anti-HBs conversion from negative (at Week 6) to positive at each scheduled visit after treatment initiation (after study Week 6), among participants who are seronegative at study Week 6
Number of participants with anti-HBe conversion from negative (at study Week 6) to positive at a subsequent visit | Entry and Weeks 6, 12, 18, 36, 54, 72, 90
  Anti-HBe conversion from negative (at Week 6) to positive at each scheduled visit after treatment initiation (after study Week 6), among participants who are seronegative at study Week 6
Change in quantitative HBeAg from pre-treatment | Entry and Weeks 6, 12, 18, 36, 54, 72, 90
  Pre-treatment value is the average of measurements at study entry and treatment initiation (study Weeks 0 and 6)
Detection of hepatitis B core-related antigen (HBcrAg) | Entry and Weeks 6, 8, 12, 14, 18, 24, 36, 54, 72,90
  Based on laboratory evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Debika Bhattacharya, MD, Study Chair — UCLA CARE Center CRS; Jordan Feld, MD, PhD, Study Chair — University Health Network / Toronto Centre for Liver Disease; Raymond T. Chung, MD, Study Chair — Massachusetts General Hospital CRS
Locations (8):
- United States (3):
  - Ucsf Hiv/Aids Crs, San Francisco, California
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - Massachusetts General Hospital CRS (MGH CRS), Boston, Massachusetts
- Brazil (2):
  - 12201, Hospital Nossa Senhora da Conceicao CRS, Porto Alegre
  - 12101, Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Rio de Janeiro
- Toronto General Hospital CRS, Toronto, Ontario, Canada
- Thailand (2):
  - Thai Red Cross AIDS Research Centre (TRC-ARC) CRS (Site # 31802), Bangkok
  - Chiang Mai University HIV Treatment (CMU HIV Treatment) CRS (Site ID: 31784), Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: * With whom?
    * Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses?
    * To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available?
    * Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://submit.mis.s-3.net/. Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data."